CLINICAL TRIAL: NCT01391364
Title: A Study to Evaluate the Product Performance of a Modified Contact Lens
Brief Title: A Study to Evaluate a Modified Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 691
Record Dates: First submitted 2011-06-16; First posted 2011-07-12 (Estimated); Results first posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Myopia
Keywords: ocular irritation
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SofLens in investigational solution (Experimental): Bausch + Lomb SofLens daily disposable contact lens packaged in an investigational storage solution.
  Interventions: Device: SofLens in investigational solution
- SofLens in currently marketed solution (Active Comparator): SofLens daily disposable contact lens packaged in currently marketed storage solution.
  Interventions: Device: SofLens in currently marketed solution

INTERVENTIONS:
Device: SofLens in investigational solution — SofLens in investigational solution, worn on a daily disposable basis for 7 days.
  Arms: SofLens in investigational solution
Device: SofLens in currently marketed solution — SofLens packaged in currently marketed solution, worn on a daily disposable basis for 7 days.
  Arms: SofLens in currently marketed solution

SUMMARY:
This study is being conducted to evaluate the product performance of SofLens daily disposable contact lenses packaged in an investigational Test solution versus SofLens daily disposable contact lenses packaged in the currently marketed solution (Control), as it relates to comfort when worn by adapted soft contact lens wearers on a daily-wear basis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be free of any anterior segment disorders.
* Subjects must be adapted lens wearers and wear a lens in each eye and each lens must be of the same manufacture and brand.
* Subjects must be myopic and require contact lens correction from -0.50 D to -6.00 D in each eye.
* Subjects must be habitual wearers of daily disposable or planned replacement (at least every 3 months) soft contact lenses.
* Subjects must live/work in an urban environment at least 6 hours per day and for at least 4 days per week throughout the duration of the study.
* Subjects must be willing and able to wear the study lenses on a daily wear basis while in an urban environment.
* Subjects living/working in the urban environment must feel challenged by harsh, drying outdoor conditions (ie dust, pollution, smog).
* Subjects must feel that being in an urban environment has a negative effect on their lens wearing experience.
* Subjects must have access to an internet connection and be able to send and receive email.

Exclusion Criteria:

* Subjects who have worn gas permeable (GP) contact lenses within the last 30 days or who have worn polymethylmethacrylate (PMMA) lenses within the last three months.
* Subjects with any systemic disease currently affecting ocular health or which in the Investigator's opinion may have an effect on ocular health during the course of the study.
* Subjects using any systemic or topical medications that will, in the Investigator's opinion, affect ocular physiology or lens performance.
* Subjects with an active ocular disease or who are using any ocular medication.
* Subjects with any grade 2 or greater finding during the slit lamp examination
* Subjects with any "Present" finding during the slit lamp examination that, in the Investigator's judgment, interferes with contact lens wear.
* Subjects with any scar or neovascularization within the central 4 mm of the cornea. Subjects with minor peripheral corneal scarring (that does not extend into the central area), that in the Investigator's judgment, does not interfere with contact lens wear, are eligible for this study.
* Subjects who are allergic to any component in the study care products.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 438 (Actual)
Dates: Start 2011-04; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Bausch & Lomb, Inc., Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 438 eligible participants (876 eyes) enrolled.
Period: Overall Study
Arm/Group | SofLens in Investigational Solution | SofLens in Currently Marketed Solution
Started | 222 | 216
Completed | 217 | 214
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Population: Demographics were reported for all dispensed, eligible participants, 222 in the investigational group and 215 in the control group.
Groups:
- Total: Total of all reporting groups
Arm/Group | SofLens in Investigational Solution | SofLens in Currently Marketed Solution | Total
Number analyzed (Participants) | 222 | 215 | 437
Age, Continuous [Mean (Full Range); unit: years] | 27.9 [18 to 40] | 27.2 [18 to 40] | 27.6 [18 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 164 | 146 | 310
  Male | 58 | 69 | 127

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes With > Grade 2 Slit Lamp Findings
Description: Graded slit lamp findings for each eye, including epithelial edema, epithelial microcysts, corneal staining, limbal and bulbar injections, upper lid tarsal conjunctival abnormalities, corneal neovascularization, and corneal infiltrates were graded for severity on a scale from 0 (No Finding) to 4 (Severe Finding). The outcome measure is any finding > grade 2, across abnormalities.
Time Frame: At 2 weeks follow up
Population: Dispensed eyes with nonmissing scores in each treatment group are included in the analysis population.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | SofLens in Investigational Solution | SofLens in Currently Marketed Solution
Number analyzed (Participants) | 218 | 215
Number analyzed (eyes) | 436 | 430
eyes | 0 | 0

2. Primary Outcome: Visual Acuity
Description: Visual acuity was assessed by distance high contrast logarithm of the minimum angle of resolution (logMAR).
Time Frame: At 2 weeks follow up
Population: Eyes assessed for visual acuity at the 2 week follow up visit are included in the analysis population.
Measure: Least Squares Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | SofLens in Investigational Solution | SofLens in Currently Marketed Solution
Number analyzed (Participants) | 203 | 200
Number analyzed (eyes) | 406 | 400
logMAR | -0.051 (0.062) | -0.046 (0.061)

3. Secondary Outcome: Symptoms and Complaints
Description: Symptoms and complaints were assessed on a scale from 0 to 100, with 0 denoting the most unfavorable symptoms/complaints. Symptoms/complaints were collected by eye from each participant and based on the participant's experience with the study lenses. Symptoms/complaints parameters included the following: Burning/stinging upon insertion, Comfort upon insertion, Overall comfort, Comfort at end of day, Ease of handling/insertion, Ease of handling/removal, Dryness, Itchiness, Redness, Vision upon insertion, Vision, Vision in low light, Lens cleanness upon insertion, Lens cleanness upon removal, and Overall impression.
Time Frame: At 2 weeks follow up
Population: Eyes assessed for symptoms/complaints at the 2 week follow up visit are included in the analysis population.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | SofLens in Investigational Solution | SofLens in Currently Marketed Solution
Number analyzed (Participants) | 217 | 213
Number analyzed (eyes) | 434 | 426
score on a scale
  Burning/stinging upon insertion | 83.2 (20.5) | 86.8 (20.5)
  Comfort upon insertion | 78.2 (20.4) | 82.7 (20.4)
  Overall comfort | 77.6 (21.0) | 79.9 (20.9)
  Comfort at end of day | 70.3 (23.8) | 70.5 (23.7)
  Ease of handling/insertion | 73.1 (24.1) | 76.3 (24.1)
  Ease of handling/removal | 87.1 (16.2) | 87.9 (16.2)
  Dryness | 74.2 (24.2) | 74.5 (24.2)
  Itchiness | 84.5 (19.1) | 87.7 (19.1)
  Redness | 86.3 (17.4) | 89.2 (17.4)
  Vision upon insertion | 86.7 (14.4) | 89.2 (14.4)
  Vision | 87.7 (14.2) | 88.7 (14.2)
  Vision in low light | 85.4 (14.6) | 86.7 (14.6)
  Lens cleanness upon insertion | 90.2 (14.2) | 91.3 (14.2)
  Lens cleanness upon removal | 84.6 (15.5) | 84.1 (15.5)
  Overall impression | 73.7 (21.2) | 75.9 (21.1)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Adverse events were not coded. Therefore, source vocabulary is not applicable. There were 444 eyes dispensed test lenses and 432 eyes dispensed control lenses, assessed for adverse events.
Arm/Group | SofLens in Investigational Solution | SofLens in Currently Marketed Solution
Serious Adverse Events (participants affected / at risk) | 0/222 | 0/216
Other Adverse Events (participants affected / at risk) | 0/222 | 0/216

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.